CLINICAL TRIAL: NCT04686578
Title: Investigation the Effect of Covid-19 Fear, Anxiety on Daily Life, Sleep Quality, and Anxiety-depression of the Patients With Fibromyalgia
Brief Title: The Effects of Covid-19 Pandemic on The Patients With Fibromyalgia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Damla Cankurtaran, Medical doctor, Diskapi Yildirim Beyazit Education and Research Hospital
Other Study IDs: Fibromyalgia-pandemi
Record Dates: First submitted 2020-12-23; First posted 2020-12-28 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Fibromyalgia; Covid-19 Fear; Covid-19 Anxiety; Daily Life; Sleep Quality; Anxiety Depression
MeSH Terms: conditions — Fibromyalgia; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fibromyalgia group: Diagnosed as Fibromyalgia according to American College of Rheumatology Fibromyalgia 2018 classification criteria over 1 year, and disease activity was stabil with the same drug at least 3 months.
- Control Group: The participants who have no physicological or severe musculoskeletal, rheumatologic diseases.

SUMMARY:
The investigators planned to analyze the effect of Covid-19 fear and anxiety on the daily life, sleep quality and depression-anxiety levels of fibromyalgia patients.

DETAILED DESCRIPTION:
Fibromyalgia; as a chronic syndrome of unknown cause with widespread body pain, fatigue, sleep disorder, cognitive impairment and anxiety. Many studies have shown a relationship between pain levels and anxiety levels in patients with fibromyalgia. Covid-19 started from Wuhan, China in December 2019 and spread worldwide. The rapid spread of this unexpected pandemic all over the world brought with it many conditions such as anxiety and stress disorders. It has been reported by experts that individuals with a predisposition to conditions such as anxiety and stress disorder in premorbidity require special attention.To evaluate the psychological effects of the Covid-19 pandemic, the Covid-19 anxiety scale was developed from Lee et al. and the Covid-19 fear scale was developed from Ahoursou et al. The investigators planned to analyzed the effect on Covid-19 fear and anxiety level on fibromyalgia patients' daily life with revised Fibromyalgia Impact questionnaire, sleep quality with Pittsburgh Sleep Quality Index, and anxiety-depression level with The Hospital Anxiety and Depression scale. This study was planned as a cross-sectional case control study.

ELIGIBILITY:
Inclusion Criteria (Fibromyalgia group):

* Patients diagnosed as Fibromyalgia syndrome according to American College of Rheumatology over 1 year
* Patients' disease activity is stabil at least 3 months Inclusion Criteria (Control group) Patients have no physicologic or severe musculoskeletal and rheumatologic diseases

Exclusion Criteria:

* Patients with having other modd disorders
* Patients with severe musculoskeletal diseases
* Patients with other rheumatologic diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Fibromyalgia group: Fifty fibromyalgia patients who met the inclusion criteria who applied to the outpatient clinic between December 2020-January 2021 and volunteered to participate in the study.
  Control Group:50 participants who will be selected from clinical staff or patients companion who meet the inclusion criteria who agree to participate in the study
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-02-15 (Estimated); Study Completion 2021-02-28 (Estimated)

PRIMARY OUTCOMES:
Level of Covid-19 anxiety | 15 seconds
  It is evaluated by the Coronavirus anxiety scale (CAS). It was developed by Lee et al. and Evren et al. were made validity and reliability of this scale in Turkish. It is 5-items scale, and each item scores between 0-4. The total score (ranging from 0 to 20) is calculated by adding up each item score. The higher the score, the greater the anxiety associated with coronavirus-19. Level of Covid-19 anxiety will be compared between fibromyalgia and control groups.
Level of Covid-19 fear | 15 seconds
  It is evaluated with The Fear Covid-19 Scale which was developed by Ahorsu et al., and it was adapted into Turkish. It is 7-item scale, each item scores with 5-pont Likert scale. Total score is 35, and the higher score describe higher fear level. Level of Covid-19 fear will be compared between fibromyalgia and control groups.

SECONDARY OUTCOMES:
The Covid-19 anxiety and fear levels on daily life the patients with fibromyalgia | 15 seconds
  The daily life of fibromyalgia patients will be analyzed with Fibromyalgia Impact questionnaire (FIQ). It has 21 individual questions. All questions are based on an 11-point numeric rating scale of 0 to 10. It is divided three domains: function, over impact, symptoms. The summed score for function (range 0 to 90) is divided by 3, the summed score or overall impact (range 0 to 20) is not changed, and the summed score for symptoms (range 0 to 100) is divided by 2. The total score is the sum of the three modified domain scores, and total score ranges from 0 to 100. Higher scores indicate worse daily life.
  Investigators will be analyzed the relationship between CAS, the fear Covid-19 Scale, and the FIQ.
The Covid-19 anxiety and fear levels on sleep quality the patients with fibromyalgia | 15 seconds
  The Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval. The sum of scores for these seven components yields one global score.The total score ranges from 0-21. A total score greater than 5 indicates "poor sleep quality" Investigators will be analyzed the relationship between CAS, the fear Covid-19 Scale, and the PSQI.
The Covid-19 anxiety and fear levels on anxiety-depression the patients with fibromyalgia | 15 seconds
  The anxiety and depression level will be evaluated with Hospital anxiety-and depression scale (HADS).The purpose of the scale is not to make a diagnosis. The scale is a self-report scale and consists of 14 questions, 7 of which investigate depression, and 7 of which investigate anxiety of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Damla Cankurtaran, MD, Principal Investigator — Diskapi Yildirim Beyazit Education and Research Hospital; Ece uNLU aKYUZ, Assoc Prof., Study Chair — Diskapi Yildirim Beyazit Education and Research Hospital; Nihal Tezel, MD, Study Chair — Diskapi Yildirim Beyazit Education and Research Hospital
Locations (1):
- Diskapi Education and Research Hospital, Ankara, Altındag, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Salameh P, Hajj A, Badro DA, Abou Selwan C, Aoun R, Sacre H. Mental Health Outcomes of the COVID-19 Pandemic and a Collapsing Economy: Perspectives from a Developing Country. Psychiatry Res. 2020 Dec;294:113520. doi: 10.1016/j.psychres.2020.113520. Epub 2020 Oct 22. PMID 33142145
- [Background] Mohabbat AB, Mohabbat NML, Wight EC. Fibromyalgia and Chronic Fatigue Syndrome in the Age of COVID-19. Mayo Clin Proc Innov Qual Outcomes. 2020 Dec;4(6):764-766. doi: 10.1016/j.mayocpiqo.2020.08.002. Epub 2020 Nov 13. No abstract available. PMID 33204998